CLINICAL TRIAL: NCT04681872
Title: Marshall Ethanolization, Pulmonary Vein Isolation and Line Completion for Ablation of Persistent Atrial Fibrillation
Acronym: MARSHALL-PLAN
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CHUBX 2019/55
Record Dates: First submitted 2020-12-18; First posted 2020-12-23 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2025-06

CONDITIONS: Atrial Fibrillation
Keywords: Persistent atrial fibrillation; Pulmonary vein isolation; Catheter ablation; Ethanolization; Ligament of Marshall
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Intervention Model Description: The Marshall Plan is a prospective randomized, parallel-group, multicenter clinical trial of superiority
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Marshall Plan arm (Experimental): Patients will undergo (1) the destruction of Marshall bundles by ethanol infusion followed by ablation of the distal coronary sinus bundles, the ridge and the saddle; (2) the standard pulmonary veins sleeves isolation; (3) and finally the ablation of the mitral, the roof, and the cavo-tricuspid isthmus.
  Interventions: Procedure: Destruction of Marshall bundles; Procedure: Pulmonary veins isolation; Procedure: Linear ablation in the left and right atria
- Pulmonary vein isolation arm (Active Comparator)
  Interventions: Procedure: Pulmonary veins isolation

INTERVENTIONS:
Procedure: Destruction of Marshall bundles — Destruction of Marshall bundles by ethanol 96% infusion (2 separate injections of 5ml on 1 minute each) followed by ablation of the distal coronary sinus bundles, the ridge and the saddle.
  Arms: Marshall Plan arm
Procedure: Pulmonary veins isolation — Achievement of a wide disconnection of the right and left pulmonary veins.
Procedure: Linear ablation in the left and right atria — Ablation of the mitral, the roof, and the cavo-tricuspid isthmus
  Arms: Marshall Plan arm

SUMMARY:
In ablation strategy for persistent Atrial Fibrillation (PsAF), ablation limited to Pulmonary Vein (PV) isolation is the most straightforward approach but the result give only 50% of arrhythmia free follow-up. Substrate modification strategies have failed to demonstrate their superiority with variable reported success rate. The Marshall network is a highly arrhythmogenic structure that has not been incorporated in current ablation strategies. The investigators sought to investigate a new ablation strategy that target systematically the vein of Marshall by ethanol infusion. This step is integrated in a new ablation strategy consisting in a global anatomical substrate based ablation including PV isolation and left atrial linear ablation (Marshall-Plan).

DETAILED DESCRIPTION:
Atrial fibrillation (AF) characterized by a fast and anarchic electrical activation of the atria, results in uncoordinated and inefficient atrial contractions that increases the risks of heart failure and strokes. Besides being a major source of morbidity and mortality, AF is one of the most common heart condition and its prevalence increases with age. Radiofrequency catheter ablation of AF has become one of the treatment of choice in AF resistant to conventional antiarrhythmic drugs. For paroxysmal AF, the ablation strategy is clear and consists in complete pulmonary veins isolation (PVI). However, if this strategy works well in paroxysmal AF, the recurrences rate remains high in persistent AF. Beyond PVI, the ablation strategy that has prevailed over the past two decades remains controversial: the left atrium partition using linear lesions ("cox-maze" strategy); the mapping of the left atrium in AF to identify and localize the arrhythmia sources. Both methods have, besides favoring atrial flutters, failed to demonstrated superiority compared to PVI alone (as showed by the clinical trial STAR AF 2). The investigators aims to test a new method of ablation for patients suffering from persistent AF in order to decrease post ablation recurrence. They propose a strategy targeting the native structures facilitating reentries including the ligament of Marshall (LOM), an embryological remnant. Indeed, two studies have demonstrated that LOM could be the source of focal activities, the substrate of reentries and a strong parasympathetic modulator. For these reasons, LOM may represent a major target in AF treatment besides PV isolation. To date, ablation techniques do not ensure the complete destruction of the Marshall's musculature and parasympathetic ganglia that surround it, largely isolated by a sheath of adipose tissue. To overcome this technical limitation, LOM elimination can be achieved by alcohol injection into the vein of Marshall. This innovative approach will then consist in 3 consecutive steps: 1) the destruction of Marshall bundles by ethanol infusion followed by the ablation of the distal and proximal muscular ramification (coronary sinus and ridge); 2) the standard PV isolation; 3) the linear lesions: the mitral, the roof and of the cavo-tricuspid isthmus, main causes of recurrence in atrial flutter.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years of both genders
* Suitable candidate for catheter and ablation of atrial fibrillation defined as: history of symptomatic persistent atrial fibrillation in the past year documented by ECG,
* Patient affiliated or beneficiary of social security scheme,
* Free, informed and written consent signed by the participant and the principal investigator (at least at the inclusion date and before all exams required for the clinical research),
* Effective contraception for women of childbearing potential.

Exclusion Criteria:

* Prior left atrial heart ablation procedure,
* Documented left atrial thrombus or another abnormality which precludes catheter introduction,
* Contraindication to anticoagulation therapy (heparin, warfarin, or novel oral anticoagulant (NOAC)),
* Contraindication to iodinated contrast products (history of major immediate reaction, thyrotoxicosis),
* Ethanol hypersensitivity,
* Unstable angina or ongoing myocardial ischemia,
* Myocardial infarction within 3 months prior to inclusion,
* Congenital heart disease, where the underlying abnormality increases the ablation risk,
* Severe bleeding, clotting or thrombotic disorder,
* Hypertrophic cardiomyopathy defined by a left ventricular septum thickness > 1.5 cm,
* Pregnant, parturient or nursing women,
* Person unable to give informed consent,
* Patient detained by judicial or administrative order, patient under legal protection (guardianship, curators, safeguarding justice).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 262 (Actual)
Dates: Start 2021-09-20 (Actual); Primary Completion 2027-09-20 (Estimated); Study Completion 2027-09-20 (Estimated)

PRIMARY OUTCOMES:
Recurrence of AF or Atrial Tachycardia (AT) greater than 30 seconds with or without antiarrhythmic medications after a single ablation procedure | 2 years
  Recurrence rate (percentage) of AF or AT > 30 seconds after the blanking period of 3-months post ablation, at 2 years with or without antiarrhythmic medications after a single ablation procedure. Recurrences will be identified through transtelephonic electrocardiogram (ECG) monitor with weekly transmitted ECG and at any time in case of symptoms.

SECONDARY OUTCOMES:
Recurrence of AF or AT greater than 30 seconds after multiple ablation procedures | 2 years
  Recurrence rate (percentage) of AF or AT > 30 seconds after the blanking period of 3-months post procedure, at 2 years after multiple ablation procedures. It will be identified through transtelephonic ECG monitor with weekly transmitted ECG and at any time in case of symptoms.
Recurrence of AF or AT greater than 30 seconds after a single ablation procedure (1) | 2 years
  Recurrence rate (percentage) of AF or AT > 30 seconds after the blanking period of 3-months post procedure, at 2 years, will be identified through transtelephonic ECG monitor with weekly transmitted ECG and at any time in case of symptoms.
Recurrence of AF greater than 30 seconds after a single ablation procedure (2) | 2 years
  Recurrence rate (percentage) of AF > 30 seconds after the blanking period of 3-months post procedure, at 2 years after a single ablation procedure. It will be identified through transtelephonic ECG monitor with weekly transmitted ECG and at any time in case of symptoms.
Recurrence of AF greater than 30 seconds after multiple ablation procedure. | 2 years
  Recurrence rate (percentage) of AF > 30 seconds after the blanking period of 3-months post procedure, at 2 years after a multiple ablation procedure. It will be identified through transtelephonic ECG monitor with weekly transmitted ECG and at any time in case of symptoms.
Recurrence of AF or AT greater than 30 seconds without antiarrhythmic medications after a single ablation procedure. | 2 years
  Recurrence rate (percentage) of AF or AT > 30 seconds after the blanking period of 3-months post procedure at 2-years without antiarrhythmic medications after a single ablation procedure. It will be identified through transtelephonic ECG monitor with weekly transmitted ECG and at any time in case of symptoms.
Recurrence of AF or AT greater than 30 seconds without antiarrhythmic medications after multiple ablation procedure. | 2 years
  Recurrence rate (percentage) of AF or AT > 30 seconds after the blanking period of 3-months post procedure at 2-years without antiarrhythmic medications after multiple ablation procedure. It will be identified through transtelephonic ECG monitor with weekly transmitted ECG and at any time in case of symptoms.
Proportion of patients under antiarrhythmic medications | 2 years
  Percentage of patients
Proportion of patients with repeated procedures | up to 2 years
  Percentage of patients
Incidence of periprocedural complications | 2 years
  Percentage of periprocedural complications : transient ischemic attack or stroke, cardiac tamponade, atrioesophageal fistula, pericarditis, complications at access site (hematoma, arteriovenous fistula, pseudoaneurysm)

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas DERVAL, MD, Principal Investigator — University Hospital, Bordeaux; Antoine BENARD, MD, Study Chair — University Hospital, Bordeaux
Locations (9):
- AZ Sint Jan Brugge, Bruges, Belgium
- France (8):
  - Clinique Saint Augustin, Bordeaux
  - Clermont-Ferrand University Hospital, Clermont-Ferrand
  - Ambroise Paré Hospital, Neuilly-sur-Seine
  - Les Franciscaines Hospital, Nîmes
  - Bordeaux University Hospital, Pessac
  - Centre Cardiologique du Nord, Saint-Denis
  - Clinique Pasteur, Toulouse
  - Toulouse University Hospirtal, Toulouse